CLINICAL TRIAL: NCT04558866
Title: Extreme Bipolar Androgen Therapy With Darolutamide and Testosterone Cypionate in Patients With Metastatic Castration-Resistant Prostate Cancer (ExBAT Trial)
Acronym: ExBAT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 0620
Record Dates: First submitted 2020-09-11; First posted 2020-09-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate; darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExBAT Arm (Experimental): Testosterone Cypionate 400 mg IM on Day 1 and Darolutamide 1,200mg/day (two 300 tablets every 12 hours) p.o. for 28 days, from day 29 to day 56 followed by a washout period of 7 days (63-day cycles), until loss of benefit (disease progression and/or limiting toxicity).
  Interventions: Drug: Testosterone Cypionate; Drug: Darolutamide

INTERVENTIONS:
Drug: Testosterone Cypionate — One administration every 63 cycles until progression or unacceptable toxicity or completion of treatment phase (54 weeks; 6 cycles), whichever comes first.
  Other Names: Deposteron
Drug: Darolutamide — During 4 weeks, from day 29 to day 56 of each 63-day cycle (+- 3 days) until progression or unacceptable toxicity or completion of treatment phase (54 weeks; 6 cycles), whichever comes first.
  Other Names: Nubeqa

SUMMARY:
This is a multi-center, open-label, phase II, single-arm trial evaluating combination of darolutamide and high testosterone doses - extreme bipolar androgen therapy (ExBAT) - in patients with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is a multi-center, open-label, phase II, single-arm trial evaluating combination of darolutamide and high testosterone doses - extreme bipolar androgen therapy (ExBAT) - in patients with metastatic castration-resistant prostate cancer (mCRPC) progressing after abiraterone. Extreme androgen therapy will include alternating 56-day cycles of darolutamide 1,200mg/day (two 300 tablets every 12 hours) p.o. for 28 days followed by testosterone cypionate 400 mg i.m. During the treatment period, patients will be followed with chest, abdomen and pelvis CT and bone scan every 8-9 weeks until cycle 4 and every 12 weeks thereafter during the study period. Patients who present with disease progression but are considered to be benefiting from the treatment may continue receiving it, but will be followed by their treating physician according to local guidelines (follow-up period). All patients who stopped treatment will enter follow-up period and survival data will be collected from medical charts. Additionally, QoL questionnaires (BPI-SF, EQ-5D-3L and FACT-P) will be applied every 8-9 weeks until the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.
2. Male aged 18 years and above.
3. Histologic confirmation of adenocarcinoma of the prostate.
4. Evidence of M1 metastatic disease (as defined by AJCC criteria) on previous bone, CT, and/or MRI scan.
5. Ongoing androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone (GnRH) analogue or bilateral orchiectomy (ie, surgical or medical castration) confirmed by testosterone level below 50 ng/dL at the screening visit. Castrate levels of testosterone must be maintained by surgical or medical means (luteinizing hormone-releasing hormone [LHRH]/ GnRH analogues) throughout the conduct of the study.
6. Documented prostate cancer progression as per PCWG3 criteria1-3 with at least one of the following:

   * PSA progression: defined by a minimum of 2 rising PSA levels with an interval of ≥ 1 week between each determination. The PSA value at the screening visit should be ≥ 2 ng/mL.* Participants who received an anti-androgen must have progression after withdrawal (4 weeks since last flutamide, bicalutamide or nilutamide administration)
   * Radiographic disease progression in soft tissue based on RECIST 1.1 criteria. Participants whose disease spread is limited to regional pelvic lymph nodes will be considered eligible.
   * Radiographic disease progression in bone defined as appearance of 2 or more new bone lesions on bone scan.
7. ECOG performance status 0-1.
8. Participants who are chemotherapy-naive for mCRPC who have received prior treatment with abiraterone acetate for advanced prostate cancer (M1 castration-sensitive or M1 castration-resistant settings). Abiraterone should be stopped at least 14 days prior to study treatment initiation.
9. Participants already receiving agents for the management of skeletal-related events (SREs) are allowed to continue with anti-bone resorptive therapy (including, but not limited to bisphosponate or receptor activator of nuclear factor kappa ligand inhibitor) if on stable dose for more than 28 days prior to treatment arm assignment.
10. Prior prostate cancer vaccine therapy, radiation therapy, radium-223, anti-androgens (eg, flutamide), ketoconazole, and diethylstilbestrol (DES) or other estrogens, are allowed up to 28 days prior to study arm assignment.
11. Asymptomatic or minimally symptomatic mCRPC according to Brief Pain Inventory - Short Form (BPI-SF) performed during screening: asymptomatic is defined as BPI-SF item #3 score of 0 to 1; minimally symptomatic is defined as BPI-SF item #3 score of 2 to 4.
12. Patients must agree to refrain from donating sperm during the course of this study and for at least 1 week after completion of study therapy.
13. Sexually active male subjects with female partners of childbearing potential must agree to use an adequate method of contraception as outlined in "Section 5.3.4 Contraception" during the course of the study treatment with Darolutamide and for 1 week after last dose.
14. Sufficient tumor tissue obtained prior to enrollment from a metastatic tumor lesion or from a primary tumor lesion (formalin fixed paraffin-embedded [FFPE] block or unstained tumor tissue sections). Tumor sample may be from core biopsy, punch biopsy, excisional biopsy, or surgical specimen). For patients without an available archival sample prior to study entry, enrolment without tissue provision will be allowed.

Exclusion Criteria:

1. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast.
2. Participants with active brain metastases. Participants with brain metastases are eligible to enroll in this study if brain metastases have been treated and there is no magnetic resonance imaging (MRI except where contraindicated in which CT scan is acceptable) evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to first dose of study drug administration.
3. Participants must have recovered from the effects of major surgery requiring general anesthesia or significant traumatic injury at least 14 days before treatment arm assignment.
4. Prior chemotherapy for mCRPC. Prior docetaxel for metastatic hormone-sensitive prostate cancer is allowed if ≥ 12 months elapsed from last dose of docetaxel.
5. Prior treatment with enzalutamide, apalutamide, darolutamide or any 2nd generation anti-androgen for prostate cancer.
6. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent or completing quality of life questionnaires.
7. Participants with serious or uncontrolled medical disorders that, in the opinion of the investigator, would impair the ability of the participant to receive protocol therapy or obscure the interpretation of AEs.
8. Patients who are unable to swallow oral medications.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. History of acute myocardial infarction (AMI), cerebrovascular accident and/or coronary artery stent or bypass surgery within 6 months of study entry.
11. Gastrointestinal disorders likely to interfere with absorption of the study medication.
12. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place.
13. Uncontrolled hypertension despite medical management as indicated by systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg at the screening visit. Patients may be re-screened after adjustments of anti- hypertensive medications.
14. Inadequate organ function and laboratory tests as follows:

    * WBC < 2.0 x 109/L; Neutrophils < 1.5 x 109/L; Platelets <100x109/L; Hemoglobin < 9.0 g/dL (no history of red blood cell transfusion within 4 weeks prior to study entry).
    * Serum creatinine > 2x ULN unless creatinine clearance ≥ 40 mL/min (measured or calculated using the Cockroft-Gault formula).
    * AST or ALT: > 3.0 x ULN; Total bilirubin >1.5 x ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0x ULN).
15. History of allergy or hypersensitivity to study drug components.
16. Any psychological, familial, sociological, or geographical condition that may hamper compliance with the protocol and follow-up.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Radiographic Progression-Free Survival (rPFS) | 12 months
  Defined as (at least one of the 3 criteria below):
  * Bone progression according to the Prostate Cancer Working Group 3 (PCWG3):
    * The first bone scan with ≥2 new lesions compared to baseline is observed <12 weeks from randomization and is confirmed by a second bone scan taken ≥6 weeks later showing ≥2 additional new lesions (a total of ≥4 new lesions compared to baseline);
    * The first bone scan with ≥2 new lesions compared to baseline is observed ≥12 weeks from randomization and the new lesions are verified on the next bone scan ≥6 weeks later (a total of ≥2 new lesions compared to baseline).
  * Progression of soft tissue lesions measured by CT or MRI as defined in modified RECIST criteria.
  * •Death from any cause. The first bone scan with ≥2 new lesions compared to baseline is observed ≥12 weeks from randomization and the new lesions are verified on the next bone scan ≥6 weeks later (a total of ≥2 new lesions compared to baseline).

SECONDARY OUTCOMES:
PSA decline ≥ 50% rate from baseline (PSA50) | 54 weeks
  Defined as a decrease in the PSA ≥ 50% compared to the baseline value, confirmed by a second measurement at least 4 weeks apart. Patients will perform PSA test on Day 1 and Day 29 of each cycle during the study.
Time to disease progression | 54 weeks
  Defined as the time from Cycle 1 Day 1 of therapy to the date of first PSA, Clinical or Radiographic progression, whichever comes first. Patients not experiencing PSA, clinical or radiographic progression as of database cut-off, whether or not surviving, will be censored at the last assessment. The PSA progression will be defined as per PCWG3 guidelines: for patients showing an initial decline in PSA from baseline, is defined as an increase in PSA that is ≥ 25% and ≥ 2 ng/mL above the nadir, and which is confirmed by a second value at least 4 weeks later (i.e. aconfirmed rising trend). For patients with no decline in PSA from baseline, is defined as an increase in PSA that is ≥ 25% and ≥ 2 ng/mL after 12 weeks.
Radiographic progression-free survival (rPFS) | 54 weeks
  Defined as the time of the first dose to objective clinical or radiographic tumor progression as defined by PCWG3 for progressive disease or death. Progression will be assigned to the earliest observed time. Patients whose disease has not progressed at follow-up will be censored at the date when the last tumor assessment determined a lack of progression.
Overall survival (OS) | 54 weeks
  Defined as the time from Cycle1 Day 1 to date of death due to any cause. Patients who are still alive or who are lost to survival follow-up as of database cut-off date will be censored at the last known alive date on or prior to database cut-off date.
Quality of life (QoL) - EQ-5D-3L | 54 weeks
  QoL will be assessed using EQ-5D 3 level version [EQ-5D-3L] questionnaire. Summary statistics of the scores will be reported at baseline, and then on Day 1 of each cycle (+- 7 days), while the patient is on the study up to 54 weeks.
Quality of life (QoL) - FACT-P | 54 weeks
  QoL will be assessed using Functional Assessment of Cancer Therapy- Prostate [FACT-P] questionnaire. Summary statistics of the scores will be reported at baseline, and then on Day 1 of each cycle (+- 7 days), while the patient is on the study up to 54 weeks.
Quality of life (QoL) - BPI-SF | 54 weeks
  QoL will be assessed using Brief Pain Inventory-Short Form [BPI-SF]) questionnaire. Summary statistics of the scores will be reported at baseline, and then on Day 1 of each cycle (+- 7 days), while the patient is on the study up to 54 weeks.
Frequency and severity of adverse events | Until 28 days after treatment discontinuation
  Incidence of adverse events (based on CTCAE Version 5) summarized by system organ class and/or preferred term, severity and relation to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Assed Bastos, Principal Investigator — Latin American Cooperative Oncology Group; Pedro Henrique Isaacson Velho, Principal Investigator — Latin American Cooperative Oncology Group
Locations (6):
- Brazil (6):
  - Hospital São Rafael - Oncologia D'Or BA, Salvador, Estado de Bahia
  - Hospital Sírio-Libanês DF, Brasília, Federal District
  - CTTB - Centro de Tratamento de Tumores Botafogo (Oncoclínicas), Rio de Janeiro, Rio de Janeiro
  - HMV - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sírio-Libanês SP, São Paulo, São Paulo
  - HIAE - Hospital Israelita Albert Einstein, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No